CLINICAL TRIAL: NCT02991924
Title: Risk Factors of Medistinal Metastasis in Endoscopic Medistinal Staging of Non-small Cell Lung Cancer
Brief Title: Risk Factors of Medistinal Metastasis in Endoscopic Staging of Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Bin Hwangbo, Principal Investigator, National Cancer Center, Korea
Other Study IDs: NCC2016-0156
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: endobronchial ultrasound; EBUS-TBNA; lung cancer; staging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate risk factors for mediastinal lymph node metastasis in potentially operable non-small cell lung cancer in order to find indications for endoscopic mediastinal staging. Chest CT, integrated PET/CT, and endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA) +/- endoscopic ultrasound with bronchoscope-guided fine needle aspiration (EUS-B-FNA) are performed for mediastinal staging. CT and PET/CT findings, histologic types and other risk factors will be analyzed. The investigators develop the prediction method for mediastinal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or strongly suspected non-small cell lung cancer (NSCLC)
* Potentially operable

Exclusion Criteria:

* M1 disease
* Inoperable T4 disease
* Mediastinal infiltration or extranodal invasion of the mediastinal lymph node visible on chest CT
* Confirmed supraclavicular lymph node metastasis
* Pancoast tumours
* T1 ground glass opacity nodule (with solid part 1<cm)
* Solid T1 (1<cm)N0 M0 by CT & PET/CT
* Inoperable patients (after evaluating medical and surgical operability)
* Patients who refused surgical treatment
* Contraindications for bronchoscopy
* Drug reaction to lidocaine, midazolam, fentanyl
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Relative risk of risk factors for mediastinal metastasis | When confirmative diagnosis are available in all subjects ;3 years
  risk factors; CT staging (N0-3), PET staging (N0-3), tumor location(central or peripheral), tumor size and histologic types of lung cancer.

SECONDARY OUTCOMES:
Diagnostic values of endoscopic staging | When confirmative diagnosis are available in all subjects ;3 years
  sensitivity, negative predictive value, accuracy
Survival | After the diagnosis ; 7 years
  survival after lung cancer treatment
Molecular test | for each subject; up to 60 days, available in all subjects ; 3 years
  EGFR, ALK etc

CONTACTS AND LOCATIONS:
Overall Officials: Bin Hwangbo, PhD, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center (NCC) Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung HS, Yoon HI, Hwangbo B, Park EY, Choi CM, Park YS, Lee K, Ji W, Park S, Lee GK, Kim TS, Kim HY, Kim MS, Lee JM. Prediction Models for Mediastinal Metastasis and Its Detection by Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration in Potentially Operable Non-Small Cell Lung Cancer: A Prospective Study. Chest. 2023 Sep;164(3):770-784. doi: 10.1016/j.chest.2023.03.041. Epub 2023 Apr 3. PMID 37019355